CLINICAL TRIAL: NCT01963754
Title: Compare Articaine 1:100.000, 4% Epinephrine, Subperiosteal With Loco-regional Anesthesia for Placing Dental Implants in Posterior Mandible - Double-Blinded Randomized Clinical Trial
Brief Title: Compare Subperiosteal and Loco-Regional Anesthesia in Posterior Mandible Dental Implant Installation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Implantology Institute (Other)
Responsible Party: Principal Investigator, Andre Chen, Msc, Implantology Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: II-03
Record Dates: First submitted 2013-10-12; First posted 2013-10-16 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Surgical Complications From Local Anesthesia; Dental Implant Failed; Anesthesia Complications; Anesthesia Morbidity
Keywords: Articaine 1:100.000; Dental Implants; Posterior mandible; Loco-regional Anesthesia; Subperiosteal Anesthesia
MeSH Terms: interventions — Dental Implants; Carticaine; Epinephrine; Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subepriosteal Articaine (Experimental): Administer Subperiosteal 1:100.000 Articaine 4% epinephrine, buccal and lingually, for Dental Implants in Posterior mandible
  Interventions: Device: Dental Implants in Posterior Mandible; Drug: Subperiosteal 1:100.000 Articaine 4% epinephrine
- Loco-regional Articaine (Active Comparator): Administer Loco-regional 1:100.000 articaine 4% epinephrine, for Dental Implants in Posterior Mandible
  Interventions: Device: Dental Implants in Posterior Mandible; Drug: Loco-regional 1:100.000 Articaine 4% epinephrine

INTERVENTIONS:
Device: Dental Implants in Posterior Mandible — Place dental implants in posterior mandible, distal from canine, according to manufacturer recommendations
  Other Names: Dental Fixtures
Drug: Subperiosteal 1:100.000 Articaine 4% epinephrine — Administration of subperiosteal anesthesia for implant placement
  Other Names: Local Anesthesia
  Arms: Subepriosteal Articaine
Drug: Loco-regional 1:100.000 Articaine 4% epinephrine — Administer loco-regional anesthesia for implant placement in posterior mandible
  Other Names: Local Anesthesia
  Arms: Loco-regional Articaine

SUMMARY:
In patients that are going to receive a dental implant in the posterior mandible (distal from canine), does the subperiosteal anesthetic technique with Articaine 1:100.000 4 % Epinephrine compared to the loco-regional one, produces the same analgesia during surgery ?

DETAILED DESCRIPTION:
Inter/Intra observer agreement will be made for administration of local subperiosteal, loco-regional anesthesia, operatory evaluation of pain and radiologic examination.

One group will receive articaine 1:100.000, 4% epinephrine subperiosteal and the other 1:100.000 4% epinephrine loco-regional for dental implant installation in posterior mandible.

The evaluation parameters will focus on intraoperatory pain, Intraoperatory anesthetic complications, anesthetic efficiency, correlation between distance from implant to inferior alveolar nerve, intraoperatory pain, post-operatory at 3 and 10 days and correlate changes, and survival rate of dental implants during and post osseointegration period.

ELIGIBILITY:
Inclusion Criteria:

* Single unit implant rehabilitation
* Maxilla and mandible
* Must accept treatment plan
* Must sign informed consent
* dental extraction performed at least 3 month prior
* Must have at least 6 mm of residual bone
* Absence of oral lesions
* keratinized tissue must be present

Exclusion Criteria:

* If smoking and/or other drug addiction is present
* If local anesthetic allergy is present
* Patient subjected to chemical or radiotherapy
* if Hepatic disease is present
* If immunodepression is present
* If Pregnancy is present
* If Diabetes is present
* If Heart disease is present

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Anesthesia efficiency | During Surgery for Dental Implant installation
  Evaluate subperiosteal vs loco-regional anesthesia for implant installation in posterior mandible.
  It will be measured by the amount (mean) of anesthesia pre and intraoperatory

SECONDARY OUTCOMES:
Intraoperatory Pain | During Surgery for Implant Installation in posterior mandible
  It will be measured with a direct measure composed by pre and post operatory questionnaires with Visual Analog Scales (VAS) to patient and by two indirect measures, one to the clinician that performed the surgery and one by an external clinic psychologist, both by means of VAS score
Intraoperatory Anesthesia Complications | During Surgery for implant installation in posterior mandible
  measure the amount of adverse effects of both types of procedure (subperiosteal vs loco-regional)
Post-Operatory Outcome Changes | Baseline (T0) 3 Days (T1) 10 Days (T2)
  measure post-operatory magnitude changes in both groups (subperiosteal vs loco-regional anesthesia) from baseline to 10 Days. It will be measured in VAS the amount of pain experienced by the patient.
Time of Surgery | During Surgical Procedure
  Measure the amount of time needed to perform dental implant installation in posterior mandible in both groups (subperiosteal Vs loco-regional)
Distance To Inferior Alveolar Nerve (IAN) | Post operative Panoramic radiograph
  measure in a panoramic (orthopantomography) the distance from the implant apex to the most coronal part of the IAN and correlate to the anesthesia efficacy and operatory pain

OTHER OUTCOMES:
Osseointegration | At 8 Weeks post-surgery
  evaluate the ability of dental implants to integrate into bone, comparison between the two groups, subperiosteal vs loco-regional)

CONTACTS AND LOCATIONS:
Overall Officials: Andre Chen, Msc, Principal Investigator — Implantology Institute; João Caramês, Phd, Study Director — Implantology Institute; Helena Francisco, Msc, Study Chair — Implantology Institute; Elena Cervino, Msc, Study Chair — Implantology Institute
Locations (1):
- Instituto de Implantologia, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No